CLINICAL TRIAL: NCT04475822
Title: An Intervention Study of Intermittent Fasting and Low Carbon Diet in Patients With Metabolic Syndrome
Brief Title: Explore the Effect of Diet Intervention on Lipid Metabolism and Body Mass Index Among the Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: The Hospital for Sick Children (Other); Leiden University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF2020LSK-003
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent fasting (Experimental): During the three-month intervention period, participants were allowed to eat for eight consecutive hours and fast for 16 hours a day.The eating time can be freely chosen in the following two periods: 8:00 -- 16:00;12:00 -- 20:00.No specific restriction shall be made on the type and quantity of food.
  Interventions: Behavioral: Intermittent fasting
- Low carb diet (Experimental): According to the definition of low carbon diet given by R. D. Feinman et al. (Nutrition, 2015), the daily carbohydrate intake of participants in this group was limited to 130g/ D, and the recommended diet was formulated according to the standard and combined with the local eating habits in Xi 'an, and dietary habit education was conducted. Participants could eat according to the recommended diet.
  Interventions: Behavioral: Low carb diet
- Low carbon diet and intermittent fasting group (Experimental): Participants fasted for 16 hours a day and ate for eight consecutive hours on the same diet as the low-carb group.
  Interventions: Behavioral: Low carbon diet and intermittent fasting group

INTERVENTIONS:
Behavioral: Intermittent fasting — Intermittent fasting group:During the three-month intervention period, participants were allowed to eat for eight consecutive hours and fast for 16 hours a day.The eating time can be freely chosen in the following two periods: 8:00 -- 16:00;12:00 -- 20:00.No specific restriction shall be made on the type and quantity of food.
  Other Names: Low carb diet; Low carbon diet and intermittent fasting group
  Arms: Intermittent fasting
Behavioral: Low carb diet — Low carb diet:The daily carbohydrate intake of participants in this group was limited to 130g/ D, and the recommended diet was formulated according to the standard and combined with the local eating habits in Xi 'an, and dietary habit education was conducted. Participants could eat according to the recommended diet.
  Arms: Low carb diet
Behavioral: Low carbon diet and intermittent fasting group — Low carbon diet and intermittent fasting group:Participants fasted for 16 hours a day and ate for eight consecutive hours on the same diet as the low-carb group.
  Arms: Low carbon diet and intermittent fasting group

SUMMARY:
The prevalence of metabolic syndrome (MetS) is increasing all over the world, which is largely related to the increasing obesity population and the current inactive lifestyle of human beings. It is a common problem facing public health and clinical practice.Metabolic syndrome is an accumulation of biologically metabolic risk factors related to cardiovascular disease and diabetes, including glucose metabolism disorders, hypertension, dyslipidemia, and obesity (especially central obesity).Researchers believe that the common pathological basis of these manifestations is insulin resistance, which is generally considered to be a reduction in the biological effects of insulin compared with the normal biological effects of expected biological phenomena.Nowadays, there are more and more studies on insulin resistance in the world. We have known that age, poor living and eating habits, high blood fat, high blood sugar and stress all lead to insulin resistance.

The researchers hope to reduce weight, reduce body fat rate, improve body fat distribution and insulin resistance, reverse abnormal metabolic indicators, and ultimately reduce the incidence of chronic diseases in patients with metabolic syndrome through the intervention of lifestyle and diet habits in the early stage of the disease.

ELIGIBILITY:
Inclusion criteria

1. Diagnosed with metabolic syndrome (i.e., more than 3 abnormal findings out of 5):

   1. Waist circumference ≥ 90 cm (men) or ≥ 80 cm (women).
   2. Elevated TG (use of medications for elevated TG is an alternate indicator) ≥ 150 mg/dL (1.7 mmol/L).
   3. Reduced HDL-c (use of medications for reduced HDL-c is an alternate indicator) < 40 mg/dL (1.0 mmol/L) in males < 50 mg/dL (1.3 mmol/L) in females.
   4. Elevated blood pressure (use of hypoglycemic medications is an alternate indicator). SBP ≥ 130 and/or DBP ≥ 85 mmHg.
   5. Elevated FBG (used of hypoglycemic medications is an alternate indicator) ≥ 100 mg/dL (5.6 mmol/L).
2. Age from 18 to 65 years.
3. Stable weight (change ≤ 10% current body weight) for 3 months prior to the study.
4. If participates were on hypoglycemic medications, hypotensive medications, lipid-lowering medications and cardiovascular medications, dose adjustment was not permitted during the 3-month intervention.

Exclusion criteria

1. Pregnant or breast-feeding.
2. Night shift workers.
3. History of major diseases or related diseases, such as inflammatory disease, rheumatologic disease, adrenal disease, malignancy, type 1 diabetes, cirrhosis, chronic kidney disease, acquired immunodeficiency syndrome, eating disorder, uncontrolled psychiatric disorder and major adverse cardiovascular event.
4. Current participate in other weight-management program, current on a prescribed diet for special disease or current on any drugs that effect appetite.
5. History of weight-loss surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
weight | Three months after the intervention
  kg
body fat | Three months after the intervention

SECONDARY OUTCOMES:
blood pressure | Three months after the intervention
  mmHg
blood glucose | Three months after the intervention
  mmol/L
blood lipid | Three months after the intervention
  mmol/L
uric acid | Three months after the intervention
  µmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Bingyin Shi, Study Chair — First Affilicated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Zheng Y, Wang J, Liu M, Zhou X, Lin X, Liang Q, Yang J, Zhang M, Chen Z, Li M, Wang Y, Sui J, Qiang W, Guo H, Shi B, He M. Time-restricted eating with or without a low-carbohydrate diet improved myocardial status and thyroid function in individuals with metabolic syndrome: secondary analysis of a randomized clinical trial. BMC Med. 2024 Sep 4;22(1):362. doi: 10.1186/s12916-024-03595-6. PMID 39227921
- [Derived] Zheng Y, Wang X, Wang J, Yang J, Wang T, Li Q, Zhu W, Wang Y, Sui J, Qiang W, Guo H, Wang Y, Shi B, He M. Effects of time-restricted eating and low-carbohydrate diet on psychosocial health and appetite in individuals with metabolic syndrome: A secondary analysis of a randomized controlled trial. Clin Nutr. 2024 Oct;43(10):2316-2324. doi: 10.1016/j.clnu.2024.08.029. Epub 2024 Aug 30. PMID 39226719
- [Derived] He M, Wang J, Liang Q, Li M, Guo H, Wang Y, Deji C, Sui J, Wang YW, Liu Y, Zheng Y, Qian B, Chen H, Ma M, Su S, Geng H, Zhou WX, Guo X, Zhu WZ, Zhang M, Chen Z, Rensen PCN, Hui CC, Wang Y, Shi B. Time-restricted eating with or without low-carbohydrate diet reduces visceral fat and improves metabolic syndrome: A randomized trial. Cell Rep Med. 2022 Oct 18;3(10):100777. doi: 10.1016/j.xcrm.2022.100777. Epub 2022 Oct 10. PMID 36220069